CLINICAL TRIAL: NCT00841581
Title: Intravitreal Lucentis (iL) (Ranibizumab) for the Treatment of AMD Related Pigment Epithelial Detachment (PED)
Brief Title: Lucentis to Treat Pigment Epithelial Detachment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Thomas G. Sheidow, Vitreoretinal Surgeon, Associate professor of Ophthalmology, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-08-410; 15392 (Other: REB)
Record Dates: First submitted 2009-02-09; First posted 2009-02-11 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Pigment Epithelial Detachment
Keywords: Age Related Macular Degeneration; Pigment Epithelial Detachment; Intravitreal Detachment; Anti-VEGF
MeSH Terms: conditions — Retinal Detachment; Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lucentis (Experimental): All patients receive iL for for first 6 months of study. At 6 months - patients are classified as "responders" or "non-responders". "Responders" receive iL PRN based on OCT,clinical exam etc. "Non-responders" are seen again at 12 months for repeat investigations.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Ranibizumab 0.5 mgs. (0.05 mls.) intravitreally for 6 months then as needed prn for 6 months.
  Other Names: Lucentis; DIN 02296810

SUMMARY:
Patients with Pigment Epithelial Detachments secondary to Age-Related Macular Degeneration (AMD) will receive intravitreal Lucentis monthly for 6 months in the hope of improving visual acuity from a baseline evaluation.

DETAILED DESCRIPTION:
Background:

Exudative Age Related Macular Degeneration (AMD) results in a significant and severe visual loss if left untreated as documented in natural history and observational arms of studies such as the macular photocoagulation study (MPS) and the Tap and VIP study with Visudyne. It is also clear however, that the different lesion types (classified by intravenous fluorescein angiography ((IVFA)) as occult, minimally classic or predominately classic) have both a different natural history and a different response to treatment.

The recent introduction of the anti-VEGF agents such as Macugen and Lucentis have significantly advanced our ability to treat AMD as both agents show clear efficacy across all lesion subtypes regardless of lesion composition.

A clear absence of literature on clinical outcomes exist however for fibrovascular pigment epithelial detachments (PED). PED represents a form of exudative AMD which clearly behaves in a unique and distinctive manner when compared to the lesion(s) described above.

As standard exclusion criteria within most of the major AMD trials, lesion composition of any IVFA subtype is acceptable as long as less then 50% of the lesion is composed of blood or pigment epithelial detachment. This has resulted in a notable absence of clinical literature on the response of predominately PED type lesions to current standard of care anti-VEGF agents. In an effort to address this absence, a prospective evaluation of the response of predominately PED type lesions to Lucentis, the current gold standard therapy is needed.

Study design:

Thirty two patients will be recruited to participate based on the Inclusion / Exclusion Criteria described in a later paragraph.

Patients will receive monthly intravitreal Lucentis injections every 33 days (+/- 4 days) for 6 months. At 6 months, patients will be evaluated based on ETDRS Visual Acuity and OCT to determine response to Lucentis therapy. Patients not experiencing a visual improvement from baseline ETDRS acuity (defined as a net gain from baseline of 10 or more letters) or showing a reduction in the height of the fibrovascular PED lesion on OCT of greater than 30% from baseline OCT will be deemed Lucentis non-responders. These patients will receive no further intravitreal Lucentis injections, but will undergo re-evaluation at 12 months.

Patients deemed responders, will continue with an OCT-guided 6 months active treatment period. In these patients, iL will be administered if evidence of visual loss of 1 or more lines (Snellen) from 6-month visit values, evidence of intraretinal or subretinal fluid on OCT, or growth of PED by greater than 50 microns from the 6-month visit OCT values.

Non-responders will be evaluated only at the 12-month final visit.

Baseline IVFA, OCT, Snellen Visual Acuity, ETDRS refraction and contrast sensitivity will be obtained along with a comprehensive ophthalmological examination. Complete diagnostic assessments including fluorescein angiography, OCT and visual function testing will be repeated at 3, 6 and 12 months after baseline treatment. In addition, patients who will continue on active intravitreal Lucentis therapy beyond 6 months (responders), will undergo monthly OCT examinations (months 6 through 11) and ophthalmic safety examinations in order to determine the need for Lucentis administration.

At the final, Month 12 visit, all patients will undergo ophthalmic examination, OCT, ETDRS refraction, Snellen Visual Acuity and contrast sensitivity.

ELIGIBILITY:
Inclusion Criteria:

1. Predominantly PED type lesions as classified on IVFA and OCT secondary to AMD.
2. PED under the geometric center of the foveal avascular zone.
3. Evidence of recent disease progression as suggested by one or more of the following: sub-retinal lipid or cystic macular edema, sub-retinal hemorrhage, vision loss within the last 3 months or documented lesion growth on FA over previous 6 months.
4. Visual acuity of between 20/40 and 20/800 in the study eye - Equivalent to Early Treatment of Diabetic Retinopathy Study (ETDRS) eye chart score of 5 to 75 letters at 2 meters.
5. Ambulatory Vision in the fellow eye
6. Willingness and ability to participate and provide written informed consent.

Exclusion Criteria:

1. Individuals with choroidal neovascularization from causes other than AMD.
2. Patients physically unable to tolerate intravenous fluorescein angiography
3. Any intraocular surgery within 2 months in the study eye.
4. Prior retinal or vitreous surgery including vitrectomy or scleral buckling in the study eye.
5. Any significant ocular disease that has compromised or could compromise vision in the study eye and confound analysis of the primary outcome.
6. Individuals with physical or mental disabilities that prevent accurate vision testing.
7. History of treatment of CNVM in the study eyes other than extrafoveal confluent laser photocoagulation.
8. Prior photodynamic therapy for CNV.
9. Any patient with recent history of new onset cardiac disease or thromboembolic CNS event in the past.
10. Women of childbearing potential who are not on two forms of effective contraception during the trial and for at least 60 days following the last dose of study medication.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-12; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To investigate whether iL given monthly for 6 months in patients with Predominantly PED lesions (secondary to AMD) will significantly improve mean visual acuity from baseline on a standardized ETDRS chart. | 6 months

SECONDARY OUTCOMES:
To evaluate the effect of iL given monthly for 6 months in patients with Predominantly PED lesions on lesion growth and activity over the study period. | 6 months
To evaluate the effect of iL given monthly for 6 months in patients with Predominantly PED lesions alone on contrast sensitivity. | 6 months
To evaluate the effect of iL given monthly for 6 months in patients with Predominantly PED lesions on central retinal thickness via Optical Coherence Tomography (OCT). | 6 months
To evaluate the effect of iL given for up to 12 months in patients with Predominantly PED lesions on lesion growth and activity over the study period. | 12 months
To evaluate the effect of iL given for up to 12 months in patients with Predominantly PED lesions on central retinal thickness via Optical Coherence Tomography (OCT). | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Sheidow, MD, Principal Investigator — Ivey Eye Institute, LOndon, Ontario, Canada
Locations (1):
- Ivey Eye Institute, London, Ontario, Canada